CLINICAL TRIAL: NCT04301375
Title: Omission of Surgery and Sentinel Lymph Node Dissection in Clinically Low-risk HER2positive Breast Cancer With High HER2 Addiction and a Complete Response Following Standard Anti- HER2-based Neoadjuvant Therapy (ELPIS Trial)
Acronym: ELPIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Garcia Cinca (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Clinical Trial Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004559-35
Record Dates: First submitted 2020-02-14; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Mammary Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental)
  Interventions: Drug: Pertuzumab and trastuzumab FDC subcutaneous; Drug: Paclitaxel; Drug: TDM1; Drug: Endocrine therapy; Procedure: Omission surgery

INTERVENTIONS:
Drug: Pertuzumab and trastuzumab FDC subcutaneous — Pertuzumab and trastuzumab FDC subcutaneous, A loading dose of 1200 mg pertuzumab and 600 mg trastuzumab followed by a maintenance dose of 600 mg pertuzumab and 600 mg; day 1 of each 3 week cycle during 5 neoadjuvant cycles and 13 adjuvant cycles if complete response
Drug: Paclitaxel — 80 mg/m2, day 1,8,15 of each 3 week cycle during 4 cycles
Drug: TDM1 — 3,6 mg/kg, 14 adjuvant cycles if not complete response
Drug: Endocrine therapy — Adjuvant endocrine therapy will be administered as per local practice and according to recognized clinical practice guidelines
Procedure: Omission surgery — Omission of surgery and sentinel lymph node dissection in patients with HER2-E and ERBB2 high breast cancer who achieving a complete response following standard anti-HER2-based neoadjuvant therapy with paclitaxel/trastuzumab/pertuzumab

SUMMARY:
This is a prospective, single arm, open-label, exploratory study in women with primary operable HER2-positive, HER2-enriched(HER2-E)/ERBB2-high breast cancer according to PAM50 intrinsic subtype and a ERBB2 pre-defined cutoff (high vs low ERBB2 expression), to evaluate the omission of surgery and sentinel lymph node dissection in patients with HER2-E and ERBB2 high breast cancer who achieving a complete response following standard anti-HER2-based neoadjuvant therapy with paclitaxel/trastuzumab/pertuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are at least 40 years of age on the day of signing the informed consent form with histologically confirmed diagnosis of breast cancer.
* A participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential as defined in protocol OR
  2. A woman of childbearing potential who agrees to follow the contraceptive guidance in protocol during the treatment period and for at least 7 months after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Histologically confirmed invasive adenocarcinoma of the breast, with all of the following characteristics:

  * HER2-positive status by local determination according to 2018 American Society of Clinical Oncology //College of American Pathologists guidelines.
  * PAM50 HER2-enriched subtype and ERBB2-high as predefined cutoff as per central determination.
  * Unifocal invasive carcinoma: only 1 invasive focus can be observed (the tumor focus containing or not containing an in situ component)
  * Tumor largest diameter ≤2 cm as defined by breast Magnetic resonance imaging.
  * No nodal involvement (i.e. cN0). Any suspicious axillary node by ultrasound must be biopsied. If the biopsy or the fine-needle aspiration is negative of tumor cells, patient is eligible.
  * No evidence of distant metastasis (M0) by routine clinical assessment.
* Patient must have known estrogen receptor and progesterone receptor status locally determined prior to study entry
* Eligible for taxane therapy
* Willingness of the patient to omit surgery if all criteria are met following neoadjuvant therapy
* Estimated life expectancy of at least 5 years irrespective of the diagnosis of breast cancer.
* Breast cancer eligible for primary surgery
* Have provided archival tumor tissue sample or newly obtained core. Formalin-fixed, paraffin embedded tissue blocks are mandatory. Available pre-treatment Formalin-fixed, paraffin embedded core biopsy evaluable for PAM50 or possibility to obtain one.
* Have an Eastern Cooperative Oncology Group performance status of 0 to 1. Evaluation of Eastern Cooperative Oncology Group is to be performed within 7 days prior to the date of allocation
* Ability and willingness to comply with study visits, treatment, testing and to comply with the protocol.
* Have adequate organ function as defined in the protocol. Specimens must be collected within 10 days prior to the start of study treatment

Exclusion Criteria:

* A woman of childbearing potential who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior anti-cancer therapy, including investigational agents, or treatment for primary invasive breast cancer.
* Known hypersensitivity to any of the excipients of trastuzumab, pertuzumab, TDM1 or paclitaxel.
* Clinical stage II, III or IV
* History of radiotherapy in the ipsilateral breast or axilla
* History of surgery of the ipsilateral axilla
* Bilateral invasive breast cancer
* Infiltrating lobular carcinoma.
* Multicentric or multifocal breast cancer, defined as the presence of two or more foci of cancer in the same or different quadrants of the same breast.
* Patients who have undergone sentinel lymph node biopsy prior to study treatment.
* Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 12 months prior to screening.
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
  * Documented cardiomyopathy.
  * Patient has a Left Ventricular Ejection Fraction < 55% at baseline as determined by Multiple Gated acquisition scan or echocardiogram.
  * Clinical significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular block (e.g. bifascicular block, Mobitz type II and third-degree atrioventricular block)
  * Long QT Syndrome or family history of idiopathic sudden death or congenital long QT syndrome or any of the following: o Risk factors for Torsades de Pointe including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure or history of clinically significant/symptomatic bradycardia
  * Corrected QT> 500 msec or conduction abnormality in the previous 12 months.
* Has an active infection requiring systemic therapy.
* Patients with a history of previous breast cancer are excluded. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission with no therapy for a minimum of 5 years are excluded. For patients with a history of other non-breast cancers within 5 years and considered of very low risk of recurrence per investigator's judgment (for example, papillary thyroid cancer treated with surgery), eligibility is to be discussed with Study Medical Monitor.
* Has a known history of Human Immunodeficiency Virus. Note: No HIV testing is required.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen reactive) or known active Hepatitis C virus (defined as Hepatitis C virus RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 7 months after the last dose of trial treatment.
* Patients currently on following medications, which cannot be interrupted 7 days prior treatment start:

  * Any prohibited medication as per trastuzumab, pertuzumab or paclitaxel label.
  * Herbal preparations/medications, dietary supplements.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
To estimate the loco-regional invasive disease-free survival of patients who achieve a complete response | 3 years
  To estimate the loco-regional invasive disease-free survival at 3-year of patients who achieve a complete response based on imaging and a stereotactic-guided vacuum-assisted breast biopsy, and omit loco-regional surgery. 3-years loco-regional invasive disease-free survival rate is defined as time from the first date of no disease (i.e., date of stereotaxic guided biopsy) to loco-regional recurrence. Loco-regional recurrence is defined as recurrence of breast cancer in the same breast parenchyma as the original primary lesion, the axilla, regional lymph nodes, chest wall and/or skin of the ipsilateral breast.

SECONDARY OUTCOMES:
To estimate the disease-free survival at 3years of patients who achieve a complete response based on imaging and a stereotaxic guided biopsy and omit loco-regional surgery following neoadjuvant chemotherapy and dual HER2 blockade. | 3 years
To estimate the disease-free survival at 5 years of patients who achieve a complete response based on imaging and a stereotaxic guided biopsy and omit loco-regional surgery following neoadjuvant chemotherapy and dual HER2 blockade. | 5 years
To estimate the disease-free survival at 3years of patients who do not achieve a complete response based on imaging following neoadjuvant chemotherapy and dual HER2 blockade | 3 years
To estimate the disease-free survival at 5 years of patients who do not achieve a complete response based on imaging following neoadjuvant chemotherapy and dual HER2 blockade | 5 years
To compare the cost in patients with and without breast cancer surgery, not only direct cost for hospitals/public health system, but also indirect cost for public system | 5 years
  Measured the cost in monetary units
To assess the effect of investigational treatment and standard treatment on patient reported outcomes | 5 years
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30), version 3; 3.2 EORTC QLQ-BR23 (breast cancer-specific questionnaire). There are all scale with a range that goes from 0 to 100 were 0 is the worst result and 100 the best.
Incidence, duration and severity of Adverse Events assessed by the NCI Common Terminology for Classification of Adverse Events version 5, including dose reductions, delays and treatment discontinuations | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain